CLINICAL TRIAL: NCT00275288
Title: "Brain Correlates Of Affect Regulation In BPD"
Brief Title: MRI Imaging in Borderline Personality Disorder
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Charles Schultz, University of Minnesota
Other Study IDs: 0407M62321
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; BPD; amygdala; facial expression response; MRI
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Normal
- Active Disease

SUMMARY:
MRI Study for females ages 18-45 with Borderline Personality Disorder(BPD): This study is a non-treatment study that involves 2 visits. Study Hypothesis:

1. To refine and pilot test functional neuroimaging paradigms to assess the amygdala response to neutral facial expressions across positive and negative emotional contexts.
2. To assess whether patients with borderline personality disorder show a heightened amygdala response to neutral facial expressions relative to healthy controls (20 female healthy controls, 20 females with borderline personality disorder).
3. To assess the relationship between individual differences in clinical ratings of personality and affective regulation, and the amygdala response to facial expressions.

DETAILED DESCRIPTION:
The first visit will be an interview assessment and will take place at the Ambulatory Research Center (ARC), Fairview University-Riverside Campus. In addition to the interview assessment, we will ask you to complete a set of questionnaires about your behavior and mood. This first visit will last approximately 2.5-3 hours. Following the interview assessment, if you are eligible for the MRI study we will contact you to schedule an MRI scan on a separate visit. This visit will last approximately 2 hours. At this visit you will have an MRI scan of your brain. Prior to the MRI scan, you will have a practice session in an MRI simulator.

ELIGIBILITY:
Inclusion Criteria:

Female subjects ages 18-45 whom meet criteria for BPD will be included in the study. The healthy controls will also be females between the ages 18-45. The healthy controls will undergo the same diagnostic and symptom evaluations as the female patients - these interview schedules will be used mainly for determining exclusion criteria.

-

Exclusion Criteria:

1. Neither borderline personality disorder subjects or healthy controls may have a history of schizophrenia, schizoaffective disorder, bipolar illness, major depression with psychotic features, Obsessive-Compulsive Disorder (OCD), Post-Traumatic Stress Disorder (PTSD), or Generalized Anxiety Disorder (GAD).
2. Patients and healthy controls may not have a serious neurologic or other metabolic disorder or any medical condition or treatment known to affect the parameters of this study.
3. Neither patients nor healthy controls will be included in the study if they are receiving a medical treatment that requires a medication that may have psychotropic effects.
4. Neither patients nor healthy controls can have any contraindications to MRI scanning such as a metal implant, a pacemaker, or a history of claustrophobia. At the Center for Magnetic Resonance Research (CMRR), we have developed a highly specific and detailed questionnaire to ensure the safety of all participants. This questionnaire is administered prior to any and all scans.
5. Pregnant women will be excluded from the study. This will be assessed by history, date of last menstrual period and urine pregnancy test if necessary.
6. Neither patients nor healthy controls who fulfill criteria for developmental deficiency will be included.
7. Healthy controls with more than two borderline personality disorder criteria will not be eligible for study. This is to reduce the possibility of healthy controls being "near misses" to the patients and diminishing the possibility of finding difference between the patients and the healthy controls.

   -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 Female subjects ages 18-45 whom meet criteria for BPD will be included in the study. 20 healthy controls will also be females between the ages 18-45.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To refine and pilot test functional neuroimaging paradigms to assess the amygdala response to neutral facial expressions across positive and negative emotional contexts. | 2 years
  1. To refine and pilot test functional neuroimaging paradigms to assess the amygdala response to neutral facial expressions across positive and negative emotional contexts.
  2. To assess whether patients with borderline personality disorder show a heightened amygdala response to neutral facial expressions relative to healthy controls (20 female healthy controls, 20 females with borderline personality disorder).
  3. To assess the relationship between individual differences in clinical ratings of personality and affective regulation, and the amygdala response to facial expressions

SECONDARY OUTCOMES:
Secondary Outcomes | 2 years
  2) To assess whether patients with borderline personality disorder show a heightened amygdala response to neutral facial expressions relative to healthy controls (20 female healthy controls, 20 females with borderline personality disorder).
  3) To assess the relationship between individual differences in clinical ratings of personality and affective regulation, and the amygdala response to facial expressions.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Thomas, PhD, Study Director — Asst Professor, Institute of Child Development
Locations (1):
- University of Minnesota, Dept of Psychiatry, Minneapolis, Minnesota, United States

REFERENCES:
- See also: Treatment and Research Advancements Nat'l Assn for BPD — http://www.tara4bpd.org/bpd.html